CLINICAL TRIAL: NCT03211988
Title: A Phase 2 Single-Arm Multicenter Study of Entinostat in Patients With Relapsed or Refractory Abdominal Neuroendocrine (NE) Tumors
Brief Title: Entinostat Neuroendocrine (NE) Tumor
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding and drug supply
Sponsor: Antonio Fojo (Other)
Responsible Party: Sponsor-Investigator, Antonio Fojo, Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAR1117
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Neuroendocrine Tumors
Keywords: abdominal; neuroendocrine tumor; columbia; relapsed; refractory
MeSH Terms: conditions — Neuroendocrine Tumors; Recurrence | interventions — entinostat

STUDY DESIGN:
Intervention Model Description: Simon 2-stage design (optimum version)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Entinostat (Other): Eligible patients will be enrolled according to Simon's two-stage design. The dose of Entinostat is 5 mg (one tablet) orally, once every week in a 28 day cycle.
  Interventions: Drug: Entinostat

INTERVENTIONS:
Drug: Entinostat — Dose is 5 mg orally every week (days 1, 8, 15, and 22) of a 28 day treatment cycle. Study drug should be taken in the morning and on an empty stomach, at least 2 hours after a meal and at least 1 hour before the next meal. Tablets should be taken whole and not crushed.
  Other Names: SNDX-275; MS-275

SUMMARY:
This is an open-label, single arm, multi-center Phase II trial of entinostat given as a 5 mg oral dose every week (days 1, 8, 15, and 22 of a 4-week cycle) in patients with relapsed or refractory abdominal neuroendocrine (NE) tumors. Patients will continue on treatment until disease progression or intolerable toxicity occurs.

DETAILED DESCRIPTION:
Neuroendocrine tumors (NETs) are derived from NE cells that reside widely in the endocrine system and other organs and comprise a heterogeneous group of neoplasms. Because NETs can arise in a broad spectrum of locations they are associated with a broad range of symptoms that may be caused by mass effects and/or by the production of hormones or biogenic amines.

Most recently, entinostat has been shown to down-regulate the number and function of two key immunosuppressive cells, myeloid derived suppressor cells (MDSCs) and regulatory T-cells (Tregs), in the tumor microenvironment thereby enhancing the activity of immune checkpoint inhibition. To date, entinostat has been investigated alone or in combination in >900 patients with cancer in clinical studies, including >600 patients with solid tumors. Entinostat as a single agent has been studied in metastatic melanoma and in combination has been studied in metastatic non-small cell lung cancer (NSCLC), breast cancer, renal cell cancer, and colon cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed stage intravenous (IV) unresectable relapsed, or unresectable refractory abdominal neuroendocrine tumor from the last biopsy available which may be the initial diagnostic biopsy.

   Relapsed disease is defined as progressive disease following systematic therapy with lanreotide or equivalent and either Sunitinib or everolimus or both. Refractory disease is defined as disease not responding to or having progressed within 1 month of the last dose of most recent systemic therapy to include lanreotide or an analog and either sunitinib or everolimus. (Note, small cell carcinoma and large cell undifferentiated neuroendocrine tumors will be excluded from this trial).
2. Eligibility for stage 2 of the study, if the extension stage is opened, will be determined by ribonucleic acid-sequencing (RNA-seq) analysis and master regulator profile of a single fresh needle biopsy specimen obtained during study screening.
3. Documented disease that is radiographically measurable.
4. Last dose of prior therapy must be > 21 days before the first dose of study drug administration. There is no upper limit to number of prior therapies. However, the patient must have recovered from acute toxicities from the most recent therapy to grade 1 or less.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (must be done within 7 days prior to study drug administration).
6. Age 18 years or older
7. Total Bilirubin ≤ 1.5 x Upper Limit of Normal (ULN) and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x ULN (results within 7 days before study drug administration), ≤5×ULN for patients with liver metastases.
8. Serum creatinine ≤ 1.5 x ULN (results within 7 days before study drug administration)
9. Absolute neutrophil counts of ≥ 1500/μL (without growth factor support), platelet counts ≥100,000/μL (without transfusion support); and hemoglobin ≥9 g/dL results within 7 days before study drug administration.
10. Patients or their legal representative must be able to read, understand, and sign a written informed consent
11. International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5×ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants and activated partial Thromboplastin Time (aPTT) ≤1.5×ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
12. If a female of childbearing potential, has a negative serum blood pregnancy test during screening and a negative urine pregnancy test within 3 days prior to receiving the first dose of study drug. If the screening serum test is done within 3 days prior to receiving the first dose of study drug, a urine test is not required. Note: Women of childbearing potential (WoCP) are any women between menarche and menopause who have not been permanently or surgically sterilized and are capable of procreation. Permanent sterilization includes hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy but excludes bilateral tubal occlusion. WoCP include non-women who have experienced menopause onset < 12 months prior to enrollment.
13. If a female of childbearing potential, willing to use 2 methods of birth control or willing to abstain from heterosexual activity for the course of the study through 120 days after the last dose of study drug.
14. If male, agrees to use an adequate method of contraception starting with the first dose of study drug through 120 days after the last dose of study drug.

Exclusion Criteria:

Patients fulfilling any of the following criteria will not be admitted into the study:

1. Patients with another active cancer (excluding basal cell carcinoma or cervical intraepithelial neoplasia (Cervical Intraepithelial Neoplasia (CIN) / cervical carcinoma in situ) or melanoma in situ)). Prior history of other cancer is allowed, as long as there is no active disease within the prior 5 years.
2. Pregnant or lactating women. Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test documented within 3 days prior to start of study drug.
3. Patients with uncontrolled intercurrent illness, active or uncontrolled infections, or a fever >38.5°C that has not been evaluated for infection up to the day of initial dosing. Patients with documented history of tumor fever are accepted provided acute or chronic infection has been excluded as possible cause of the fever.
4. Patients who have been treated with any investigational drug within 28 days prior to the first dose of study medication, or who are receiving concurrent treatment with other experimental drugs or anti-cancer therapy.
5. Prior treatment with histone deacetylase (HDAC) inhibitors (e.g. valproic acid, Zolinza® (SAHA), romidepsin (Istodax®).
6. History of pericarditis or pericardial effusion that had required medical or surgical intervention in the last 6 months, or myocardial infarction or arterial thromboembolic events within 6 months, or experiencing severe or unstable angina, or New York Heart Association (NYHA) Class III or IV disease, or a corrected QT (QTc) interval >0.47 seconds
7. Known human immunodeficiency virus (HIV) or a history of active Hepatitis B or C as evidenced by laboratory abnormalities in addition to positive serology. Testing is not required for patients not suspected of having these conditions
8. Any condition (e.g., known or suspected poor compliance, psychological instability, geographical location, etc) that, in the judgment of the investigator, may affect the patient's ability to sign the informed consent and comply with study procedures
9. Any condition that will put the patient at undue risk or discomfort as a result of adherence to study procedures
10. Presence or history of brain metastases.
11. Uncontrolled hypertension or diabetes mellitus
12. Any contraindication to oral agents or significant nausea and vomiting, malabsorption, or significant small bowel resection that, in the opinion of the investigator, would preclude adequate absorption.
13. Allergy to benzamide or inactive components of entinostat.
14. Patients may not be taking any corticosteroid for any reason while on study and all corticosteroids must be stopped two weeks prior to initiation of study drug.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-12-23 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to Two Years
  Percentage of patients who experience a tumor size reduction from the time of initial response to tumor progression.

SECONDARY OUTCOMES:
Duration of Progression-Free Survival (PFS) | Up to Two Years
  Time from study enrollment until disease progression or death.
Duration of Overall Survival (OS) | Up to Two Years
  The length of time from either the date of diagnosis or start of treatment that years patients diagnosed with the disease are still alive.
Duration of Response for Patients who Achieve Complete Response (CR) or Partial Response (PR) | Up to Two Years
  Time from documentation of tumor response to disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Fojo, MD, PhD, Principal Investigator — Columbia University/Herbert Irving Cancer Center
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jamison JK, Zhou M, Gelmann EP, Luk L, Bates SE, Califano A, Fojo T. Entinostat in patients with relapsed or refractory abdominal neuroendocrine tumors. Oncologist. 2024 Sep 6;29(9):817-e1213. doi: 10.1093/oncolo/oyae118. PMID 38886159